CLINICAL TRIAL: NCT00808119
Title: A Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single, Escalating Oral Doses of RTI-336 in Healthy, Male Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single, Escalating Oral Doses of RTI-336 in Healthy, Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Dr. Bradford B. Walters, MD, PhD, MBA / Chief Medical Officer, RTI International
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RTI-336-001
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — 3beta-(4-chlorophenyl) tropane-2beta-(3-(4'-methylphenyl) isoxazol-5-yl) hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: RTI-336 (CTDP 31862) — The RTI-336 drug product is formulated as hard, white, gelatin capsules. The dosage levels are 0.3, 1.0, and 3.0 mg (Cohort 1) and 6.0, 12.0, and 20.0 mg (Cohort 2). Subjects will receive a single dose of the study drug on study day 1.

SUMMARY:
This is the first study to be conducted in humans for RTI-336, a new chemical entity, with evaluations focusing on the safety, tolerability, and pharmacokinetics of RTI-336 following administration of single, oral doses. RTI-336 is a novel dopamine transporter inhibitor of the 3-phenyltropane class, and is currently being developed by RTI International as a potential pharmacotherapy to treat cocaine dependence. Data from this study will be used to plan and define dose ranges for subsequent studies.

DETAILED DESCRIPTION:
Cocaine abuse has been an epidemic in the United States since the mid- to late-1970s. It is hypothesized that a medication to treat cocaine addiction should have some, but not all, of the behavioral pharmacological properties of cocaine. Substantial evidence links the euphoric highs and addictive properties of cocaine to the inhibition of the dopamine transporter (DAT) in the brain. Cocaine binds quickly and potently to this transporter and blocks the presynaptic uptake of dopamine, resulting in subjective highs and reinforcing effects in both preclinical studies and humans. Compounds that mimic the DAT-binding properties of cocaine that are less stimulating and act with a slower receptor onset and offset may prove useful as treatment for cocaine dependence. The 3-phenyltropane analog, RTI-336, is a potent and selective DAT inhibitor that has demonstrated desirable pharmacological properties in preclinical species and is an appropriate compound to test for its potential as a medication to treat cocaine dependence.

This is the first study to be conducted in humans for RTI-336, a new chemical entity, with evaluations focusing on the safety, tolerability, and pharmacokinetics of RTI-336 following administration of single, oral doses, with the possibility of identifying the maximum tolerated dose in humans. Data from this study will be used to plan for and define dose ranges for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria are met:

1. Subject provides signed and dated, written informed consent prior to any study-specific procedures being performed, including washout of any medications and compliance with food/beverage restrictions.
2. Subject is a healthy adult male, 18-50 years of age, inclusive, at the time of consent, with body weight greater than or equal to 50 kg and a body mass index (BMI) in the range of 18-30 kg/m2, where BMI = weight (kg)/[height (m)]2.
3. Subject has a negative pre-study urine drug screen and no history of cocaine use or use of other illicit drugs or substances of abuse within 12 months of the screening visit. Drugs or substances analyzed in the urine screen include cocaine, amphetamines, barbiturates, opioids, cannabinoids, benzodiazepines, phencyclidine, alcohol, and cotinine.
4. Subject is a non-tobacco user or a prior user who quit using tobacco at least 90 days prior to screening.
5. Subject has no history of any cardiovascular disease and has a normal ECG and serum troponin at screening.
6. Subject is negative for hepatitis C antibodies, hepatitis B surface antigen and human immunodeficiency virus (HIV) at screening.
7. Subject is in good general health, in the opinion of the Investigator, and as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory tests at screening. Additionally, the subject's clinical laboratory test results must meet the following criteria: Within normal limits for sodium, protein, total WBC, hematocrit, hemoglobin, reticulocyte count, platelets, AST (SGOT), ALT (SGPT), GGT, and troponin I. Within upper limit of normal and no more than 10% below lower limit: BUN creatinine, bilirubin, total alkaline phosphatase, creatine kinase, and LDH. Within 10% of normal range and considered to be not clinically significant:calcium chloride, phosphorus, albumin, globulin, cholesterol, triglycerides, and RBC. No clinically significant abnormalities: glucose, potassium, white blood cell differential, red blood cell indices, uric acid, and urinalysis.
8. Subject is willing to use barrier contraception with spermicide during sexual intercourse while enrolled in this study and for at least 30 days after the last dose of study drug.
9. Subject is willing and able to comply with study instructions and restrictions, and is available to complete the study assessments as required by the protocol.
10. Subjects is fluent in either English or Spanish

Exclusion Criteria:

A subject will be excluded from participation in the study if any of the following criteria applies:

1. Subject self-reports a history of chronic illicit drug use or chronic use of other substances of abuse.
2. Subject has a positive urine drug/alcohol/cotinine test at screening or prior to dosing in any dose period.
3. Subject has a history or evidence of hepatic, gastrointestinal, renal, respiratory, ophthalmic, cardiovascular, hematologic, endocrine/metabolic, neurologic, immunologic, oncologic or psychiatric illness or significant abnormalities.
4. Subject has a history of and/or current major depression, psychotic symptoms, or anxiety disorder(s) based on the Major Depressive Episode, Psychotic, and Anxiety Disorder modules of the Structured Clinical Interview for DSM Disorders (details documented in study protocol).
5. Subject has a family history of psychiatric illness (psychosis, depression, anxiety disorders).
6. Subject has an abnormal ECG at screening or prior to dosing in each dose period. Premature atrial contraction or premature ventricular contraction is considered abnormal, as are bundle branch blocks, second or third degree heart block, or any arrhythmia other than respiratory sinus arrhythmia. Abnormalities also include but are not limited to the following: Heart Rate < 45 or > 100 bpm; PR interval < 120 or > 220 msec; QRS duration < 70 or > 120 msec; and QTC interval (Bazett) > 460 msec.
7. Subject has a history or family history of QT prolongation, arrhythmia, or uncontrolled hypertension.
8. Subject has a history of seizure, head injury, neurosurgery or brain trauma, or a family history of non-traumatic seizure.
9. Subject is positive for hepatitis C antibodies at screening, or hepatitis B surface antigen or HIV at screening.
10. Subject has an infection of any type or clinically significant abnormality identified by the screening medical or laboratory evaluations.
11. Subject has a history of using tobacco-containing products within 90 days of screening.
12. Subject has a history of significant alcohol consumption, defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units, with 1 unit equivalent to a half-pint (220 mL) of beer, or 1 measure of spirits, or 1 glass (125 mL) of wine.
13. Subject has consumed grapefruit or grapefruit-containing, or poppy-seed or quinine-containing substances within 14 days of the first dose period.
14. Subject has used any other drug, including prescription or non-prescription medications and herbal supplements, within 30 days prior to the first dose of study drug, with the exception of acetaminophen, which may be taken up to 24 hours prior to dosing in each dose period.
15. Subject has a history or presence of gastrointestinal, hepatic or renal disease, or other condition/surgical intervention known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
16. Subject has had any acute gastrointestinal illness or infection within 2 weeks prior to first dose of study drug.
17. Subject has participated in an investigational trial within 45 days prior to the first dose of study drug.
18. Subject is unable to donate blood, has a clotting disorder(s), or has donated/lost >500 mL blood within 8 weeks prior to screening.
19. Subject has an unexplained weight loss or gain >10% within 30 days prior to screening.
20. Subject has an allergy to 3-phenyltropane analogs (e.g., brasofensine, tesofensine), heparin, haloperidol, dopamine agonists, or related compounds.
21. Subject is unable to respond to or recognize potential side effects of the study drug. This may include, but is not limited to, subjects with a mental illness or disorder.
22. Subject has any condition or set of circumstances not otherwise excluded which in the judgment of the Investigator could interfere with the subject's ability to comply with the protocol requirements and restrictions and completion of study evaluations, or could pose safety risks to the subject.
23. Subject has performed strenuous exercise within 48 hours prior to the screening examination or refuses to abstain from strenuous exercise for 48 hours prior to and 48 hours after each dose period, 48 hours prior to the day 8 visit, or 48 hours prior to the follow-up visit.
24. Subject has a screening serum troponin result above the clinical laboratory's normal range.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of RTI-336; clinical signs and symptoms, adverse events (AEs), vital signs, electrocardiographic (ECG) parameters, clinical laboratory test results | Days 0 (Baseline), 1-3, and 8

SECONDARY OUTCOMES:
Pharmacokinetic parameters of RTI-336 and metabolites | 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, and 48 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: William A. Gerson, DO, CPI, Principal Investigator — Comprehensive Phase One
Locations (1):
- Comprehensive Phase One, Miramar, Florida, United States

REFERENCES:
- [Derived] Carroll FI, Kosten TR, Buda JJ, Wang L, Walters BB. A Double-Blind, Placebo-Controlled Trial Demonstrating the Safety, Tolerability, and Pharmacokinetics of Single, Escalating Oral Doses of RTI-336. Front Pharmacol. 2018 Jul 10;9:712. doi: 10.3389/fphar.2018.00712. eCollection 2018. PMID 30042675